CLINICAL TRIAL: NCT02421588
Title: Phase III Randomized Clinical Trial of Lurbinectedin (PM01183) Versus Pegylated Liposomal Doxorubicin or Topotecan in Patients With Platinum-resistant Ovarian Cancer (CORAIL Trial)
Brief Title: Clinical Trial of Lurbinectedin (PM01183) in Platinum Resistant Ovarian Cancer Patients
Acronym: CORAIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-C-004-14
Record Dates: First submitted 2015-04-10; First posted 2015-04-20 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — PM 01183; liposomal doxorubicin; Topotecan

ARMS (2):
- Arm A (Experimental): lurbinectedin (PM01183)
  Interventions: Drug: Lurbinectedin (PM01183)
- Arm B (Active Comparator): pegylated liposomal doxorubicin
  OR
  topotecan
  Interventions: Drug: Pegylated liposomal doxorubicin (PLD); Drug: Topotecan

INTERVENTIONS:
Drug: Lurbinectedin (PM01183)
  Arms: Arm A
Drug: Pegylated liposomal doxorubicin (PLD)
  Arms: Arm B
Drug: Topotecan
  Arms: Arm B

SUMMARY:
Multicenter, open-label, randomized, controlled phase III clinical trial to evaluate the activity and safety of PM01183 versus PLD or topotecan as control arm in patients with platinum-resistant ovarian cancer. PM01183 will be explored as single agent in the experimental arm (Arm A) versus PLD or topotecan in the control arm (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Confirmed diagnosis of unresectable epithelial ovarian, fallopian tube or primary peritoneal cancer.
* Platinum-resistant disease (PFI: 1-6 months after last platinum-containing chemotherapy).
* Evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria
* No more than three prior systemic chemotherapy regimens
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) (ECOG PS) ≤ 2
* Adequate hematological, renal, metabolic and hepatic function

Exclusion Criteria:

* Concomitant diseases/conditions: cardiac disease, immunodeficiency, chronic active hepatitis or cirrhosis, uncontrolled infection, bowel obstruction, any other major illness
* Prior treatment with PM01183, trabectedin, or with both PLD and topotecan.
* Requirement of permanent or frequent (i.e., once per week) external drainages within two weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2015-05; Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - 1112, Peoria, Arizona
  - 1102, Greenbrae, California
  - 1103, La Jolla, California
  - 1116, Los Angeles, California
  - 1120, Los Angeles, California
  - 1113, Palo Alto, California
  - 1111, San Francisco, California
  - 1122, Santa Maria, California
  - 1123, West Hills, California
  - 1109, Augusta, Georgia
  - 1104, Indianapolis, Indiana
  - 1110, Covington, Louisiana
  - 1124, Scarborough, Maine
  - 1121, Brick, New Jersey
  - 1127, Albany, New York
  - 1105, New York, New York
  - 1117, Asheville, North Carolina
  - 1101, Charlotte, North Carolina
  - 1125, Charlotte, North Carolina
  - 1108, Durham, North Carolina
  - 1107, Columbus, Ohio
  - 1118, Dayton, Ohio
  - 1119, Pittsburgh, Pennsylvania
  - 1115, Greenville, South Carolina
  - 1129, Nashville, Tennessee
  - 1131, Fort Worth, Texas
  - 1128, Houston, Texas
  - 1106, Charlottesville, Virginia

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Gaillard S, Oaknin A, Ray-Coquard I, Vergote I, Scambia G, Colombo N, Fernandez C, Alfaro V, Kahatt C, Nieto A, Zeaiter A, Aracil M, Vidal L, Pardo-Burdalo B, Papai Z, Kristeleit R, O'Malley DM, Benjamin I, Pautier P, Lorusso D. Lurbinectedin versus pegylated liposomal doxorubicin or topotecan in patients with platinum-resistant ovarian cancer: A multicenter, randomized, controlled, open-label phase 3 study (CORAIL). Gynecol Oncol. 2021 Nov;163(2):237-245. doi: 10.1016/j.ygyno.2021.08.032. Epub 2021 Sep 11. PMID 34521554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First randomization/first study treatment administration took place on 26JUN2015. The cutoff date for results was 12OCT2018. 534 patients were screened; 442 were randomized at 83 sites/12 countries. 10 patients did not receive the study treatment.
Pre-assignment Details: IC;Age≥18 years;confirmed diagnosis of unresectable epithelial ovarian, fallopian tube or primary peritoneal cancer;Platinum-resistant disease;ECOG PS≤2;Adequate hematological, renal, metabolic, and hepatic function
Groups:
- Lurbinectedin: 3.2 mg/m2 i.v. as a 1-hour infusion on Day 1 q3wk (three weeks = one treatment cycle) through peripheral or central lines. A minimum total volume of 100 mL, diluted in 5% glucose or 0.9% sodium chloride solution for infusion, had to be used for administration through a central venous catheter; if a peripheral venous catheter was used, the minimum volume was 250 mL
- Control (PLD or Topotecan): Patients randomized to the Control arm were assigned to receive PLD if they had previously been treated with topotecan, or to receive topotecan if they had previously been treated with PLD. However, if the number of patients randomized to either PLD or topotecan reached 60% (i.e., 126 patients) of the total number of patients expected in the Control Arm, then the treatment of choice in the Control Arm would be restricted to the less frequent control drug until the end of accrual
Period: Overall Study
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Started | 221 | 221
Completed | 0 | 0
Not Completed | 221 | 221
Not completed — Non-treatment-related AE | 8 | 8
Not completed — Progressive disease | 152 | 135
Not completed — Death | 11 | 3
Not completed — Physician Decision | 8 | 17
Not completed — Other reason not specified | 3 | 1
Not completed — Symptomatic deterioration | 13 | 19
Not completed — Treatment-related AE | 10 | 14
Not completed — Withdrawal by Subject | 14 | 16
Not completed — Not treated | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurbinectedin | Control (PLD or Topotecan) | Total
Number analyzed (Participants) | 221 | 221 | 442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 141 | 267
  >=65 years | 95 | 80 | 175
Age, Continuous [Median (Full Range); unit: years] | 63.0 [25 to 85] | 59.0 [28 to 87] | 61.0 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 221 | 442
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 192 | 201 | 393
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 14 | 35
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79
  Romania | 11 | 11 | 22
  Spain | 40 | 46 | 86
  United Kingdom | 17 | 14 | 31
  Austria | 3 | 4 | 7
  Belgium | 21 | 19 | 40
  Bulgaria | 5 | 5 | 10
  Czechia | 5 | 5 | 10
  France | 19 | 12 | 31
  Hungary | 9 | 14 | 23
  Italy | 47 | 47 | 94
  Serbia | 5 | 4 | 9
Body mass index [Count of Participants; unit: Participants]
  ≤20 kg/m^2 | 26 | 37 | 63
  20-25 kg/m^2 | 82 | 84 | 166
  25-30 kg/m^2 | 62 | 51 | 113
  >30 kg/m^2 | 50 | 49 | 99
  Unknown | 1 | 0 | 1
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 126 | 123 | 249
    PS 1 | 87 | 94 | 181
    PS 2 | 8 | 4 | 12
Primary site [Count of Participants; unit: Participants]
  Ovarian | 196 | 195 | 391
  Fallopian | 11 | 13 | 24
  Peritoneal | 14 | 13 | 27
Histology type [Count of Participants; unit: Participants]
  Serous/Papillary | 181 | 199 | 380
  Endometrioid | 14 | 6 | 20
  Clear cell | 10 | 12 | 22
  Mucinous | 3 | 1 | 4
  Other | 13 | 3 | 16
Histologic grade [Count of Participants; unit: Participants]
  Well differentiated | 16 | 15 | 31
  Moderately differentiated | 21 | 24 | 45
  Poorly differentiated/Undifferentiated | 154 | 143 | 297
  Unknown | 30 | 39 | 69
BRCA status [Count of Participants; unit: Participants]
  BRCA1 | 10 | 8 | 18
  BRCA2 | 4 | 3 | 7
  Not mutated | 64 | 61 | 125
  Unknown | 143 | 149 | 292
Intestinal sub-occlusion [Count of Participants; unit: Participants]
  Yes | 9 | 10 | 19
  No | 212 | 211 | 423
Clinically evident ascites [Count of Participants; unit: Participants]
  Yes | 35 | 39 | 74
  No | 186 | 182 | 368
Radiological presence of ascites [Count of Participants; unit: Participants]
  Yes | 59 | 71 | 130
  No | 162 | 150 | 312
Prior radiotherapy [Count of Participants; unit: Participants]
  Yes | 6 | 5 | 11
  No | 215 | 216 | 431
Prior Cytoreductive surgery [Count of Participants; unit: Participants]
  Yes | 198 | 204 | 402
  No | 23 | 17 | 40
Other prior surgical procedures [Count of Participants; unit: Participants]
  Yes | 86 | 81 | 167
  No | 135 | 140 | 275
Weight [Median (Full Range); unit: Kg] | 65.8 [37.0 to 125.0] | 63.0 [39.0 to 142.8] | 64.4 [37.0 to 142.8]
Height [Median (Full Range); unit: cm] | 161.0 [147 to 177] | 161.0 [144 to 183] | 161.0 [144 to 183]
Body Surface Area [Median (Full Range); unit: m^2] | 1.7 [1.3 to 2.4] | 1.7 [1.3 to 2.4] | 1.7 [1.3 to 2.4]
Body mass index [Median (Full Range); unit: kg/m^2] | 25.1 [15.0 to 47.9] | 24.7 [14.5 to 56.5] | 24.9 [14.5 to 56.5]
First diagnosis to randomization [Median (Full Range); unit: months] | 23.4 [7 to 294] | 20.7 [4 to 184] | 22.05 [4 to 294]
Sites involved [Median (Full Range); unit: number of sites] | 2.0 [1 to 5] | 2.0 [1 to 7] | 2.0 [1 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival by Independent Review Committee
Description: The primary endpoint was PFS by IRC assessment, defined as the time from the date of randomization to the date of documented progression per RECIST v.1.1 or death (regardless of the cause of death). If the patient received further antitumor therapy or was lost to follow-up before PD, PFS was censored at the date of last tumor assessment before the date of subsequent antitumor treatment.
Time Frame: Time from the date of randomization to the date of PD, death (of any cause), or last tumor evaluation, whichever came first, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 221 | 221
months | 3.5 [2.1 to 3.7] | 3.6 [2.7 to 3.8]
Statistical Analysis 1: Comparison: Lurbinectedin vs Control (PLD or Topotecan); PFS between treatments; Test type: Superiority; p = 0.6294, Log Rank; Hazard Ratio (HR) = 1.057, 95% CI 2-sided [0.854 to 1.309]
Statistical Analysis 2: Comparison: Lurbinectedin; PFS (%) at 6 months; Test type: Superiority; PFS at 6 months = 24.3, 95% CI 2-sided [18.4 to 30.7] — Percent of Participants
Statistical Analysis 3: Comparison: Control (PLD or Topotecan); PFS (%) at 6 months; Test type: Superiority; PFS at 6 months = 27.5, 95% CI 2-sided [20.9 to 34.4] — Percent of Participants
Statistical Analysis 4: Comparison: Lurbinectedin vs Control (PLD or Topotecan); PFS (%) at 6 months between treatments; Test type: Superiority; p = 0.5032, Normal approximation
Statistical Analysis 5: Comparison: Lurbinectedin; PFS (%) at 12 months; Test type: Superiority; PFS at 12 months = 8.3, 95% CI 2-sided [4.7 to 13.3] — Percent of Participants
Statistical Analysis 6: Comparison: Control (PLD or Topotecan); PFS (%) at 12 months; Test type: Superiority; PFS at 12 months = 7.0, 95% CI 2-sided [3.3 to 12.5] — Percent of Participants
Statistical Analysis 7: Comparison: Lurbinectedin vs Control (PLD or Topotecan); PFS (%) at 12 months between treatments; Test type: Superiority; p = 0.6742, Normal approximation

2. Secondary Outcome: Progression-free Survival by Investigator's Assessment
Description: The primary endpoint was PFS by Investigator's Assessment, defined as the time from the date of randomization to the date of documented progression per RECIST v.1.1 or death (regardless of the cause of death). If the patient received further antitumor therapy or was lost to follow-up before PD, PFS was censored at the date of last tumor assessment before the date of subsequent antitumor treatment.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 221 | 221
months | 3.7 [3.6 to 3.9] | 3.7 [3.5 to 4.0]
Statistical Analysis 1: Comparison: Lurbinectedin vs Control (PLD or Topotecan); PFS between treatments; Test type: Superiority; p = 0.7673, Log Rank; Hazard Ratio (HR) = 0.987, 95% CI 2-sided [0.805 to 1.209]
Statistical Analysis 2: Comparison: Lurbinectedin; PFS (%) at 6 months; Test type: Superiority; PFS at 6 months = 29.0, 95% CI 2-sided [22.8 to 35.4] — Percent of Participants
Statistical Analysis 3: Comparison: Control (PLD or Topotecan); PFS (%) at 6 months; Test type: Superiority; PFS at 6 months = 27.4, 95% CI 2-sided [21.3 to 33.9] — Percent of Participants
Statistical Analysis 4: Comparison: Lurbinectedin vs Control (PLD or Topotecan); PFS (%) at 6 months between treatments; Test type: Superiority; p = 0.7385, Normal approximation
Statistical Analysis 5: Comparison: Lurbinectedin; PFS (%) at 12 months; Test type: Superiority; PFS (%) at 12 months = 8.2, 95% CI 2-sided [4.8 to 12.7] — Percent of Participants
Statistical Analysis 6: Comparison: Control (PLD or Topotecan); PFS (%) at 12 months; Test type: Superiority; PFS (%) at 12 months = 7.5, 95% CI 2-sided [4.2 to 12.2] — Percent of Participants
Statistical Analysis 7: Comparison: Lurbinectedin vs Control (PLD or Topotecan); PFS (%) at 12 months between treatments; Test type: Superiority; p = 0.8245, Normal approximation

3. Secondary Outcome: Overall Survival (OS)
Description: Calculated from the date of randomization to the date of death (death event) or last contact (in this case, survival was censored on that date).
Time Frame: From the date of randomization to the date of death or last contact, up to 12 months after last patient inclusion, for a maximum of up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 221 | 221
months | 11.4 [9.0 to 14.2] | 10.9 [9.3 to 12.5]
Statistical Analysis 1: Comparison: Lurbinectedin vs Control (PLD or Topotecan); OS between treatments; Test type: Superiority; p = 0.8021, Log Rank; Hazard Ratio (HR) = 0.956, 95% CI 2-sided [0.772 to 1.183]
Statistical Analysis 2: Comparison: Lurbinectedin; OS (%) at 12 months; Test type: Superiority; OS at 12 months = 48.2, 95% CI 2-sided [41.3 to 54.8] — Percent of Participants
Statistical Analysis 3: Comparison: Control (PLD or Topotecan); OS (%) at 12 months; Test type: Superiority; OS (%) at 12 months = 45.3, 95% CI 2-sided [38.4 to 52.0] — Percent of Participants
Statistical Analysis 4: Comparison: Lurbinectedin vs Control (PLD or Topotecan); OS (%) at 12 months between treatments; Test type: Superiority; p = 0.5515, Normal approximation
Statistical Analysis 5: Comparison: Lurbinectedin; OS (%) at 24 months; Test type: Superiority; OS (%) at 24 months = 22.3, 95% CI 2-sided [16.8 to 28.2] — Percent of Participants
Statistical Analysis 6: Comparison: Control (PLD or Topotecan); OS (%) at 24 months; Test type: Superiority; OS (%) at 24 months = 22.7, 95% CI 2-sided [17.1 to 28.7] — Percent of Participants
Statistical Analysis 7: Comparison: Lurbinectedin vs Control (PLD or Topotecan); OS (%) at 24 months between treatments; Test type: Superiority; p = 0.9253, Normal approximation

4. Secondary Outcome: Overall Response Rate (ORR) by Independent Review Committee
Description: Best antitumor response defined as the best response obtained according to RECIST v.1.1. Tumor assessment were performed at baseline and every 8 weeks from randomization until evidence of PD. Patients who discontinued treatment without PD continued with assessments.
  Antitumor activity was assessed using the RECIST v.1.1 by the appropriate method [computed tomography scan or magnetic resonance imaging]: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters; Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum; Overall Response (OR)=CR+PR.
Time Frame: At baseline and every eight weeks from randomization until evidence of PD, assessed up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 221 | 221
Participants
  Complete response | 3 | 3
  Partial response | 29 | 25
  Stable disease | 90 | 97
  Progressive disease | 83 | 72
  Unknown | 16 | 24
Statistical Analysis 1: Comparison: Lurbinectedin; Overall response rate; Test type: Superiority; ORR = 14.5, 95% CI 2-sided [10.1 to 19.8] — Percent of Participants
Statistical Analysis 2: Comparison: Control (PLD or Topotecan); Overall response rate; Test type: Superiority; ORR = 12.7, 95% CI 2-sided [8.6 to 17.8] — Percent of Participants
Statistical Analysis 3: Comparison: Lurbinectedin vs Control (PLD or Topotecan); Overall response rate between treatments; Test type: Superiority; p = 0.6772, Fisher Exact

5. Secondary Outcome: Overall Response Rate by Investigator's Assessment
Description: as for outcome 4
Time Frame: At baseline and every eight weeks from randomization until evidence of PD, assessed up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 221 | 221
Participants
  Complete response | 3 | 2
  Partial response | 32 | 35
  Stable disease | 107 | 94
  Progressive disease | 63 | 68
  Unknown | 16 | 22
Statistical Analysis 1: Comparison: Lurbinectedin; Overall response rate (ORR); Test type: Superiority; ORR = 15.8, 95% CI 2-sided [11.3 to 21.3] — Percent of Participants
Statistical Analysis 2: Comparison: Control (PLD or Topotecan); Overall response rate (ORR); Test type: Superiority; Overall response rate (ORR) = 16.7, 95% CI 2-sided [12.1 to 22.3] — Percent of Participants
Statistical Analysis 3: Comparison: Lurbinectedin vs Control (PLD or Topotecan); Overall response rate (ORR) between treatments; Test type: Superiority; p = 0.8976, Fisher Exact

6. Secondary Outcome: Duration of Response by Independent Review Committee
Description: Duration of response (DR): calculated from the date of first documentation of response per RECIST v.1.1 (CR or PR, whichever came first) to the date of documented PD or death. The censoring rules defined above for PFS were used for duration of response.
  Best antitumor response defined as the best response obtained according to RECIST v.1.1. Tumor assessment were performed at baseline and every 8 weeks from randomization until evidence of PD. Patients who discontinued treatment without PD continued with assessments.
  Antitumor activity was assessed using the RECIST v.1.1 by the appropriate method [computed tomography scan or magnetic resonance imaging]: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)=CR+PR.
Time Frame: The time from the date when the response criteria (PR or CR, whichever was reached first) were fulfilled, to the first date when PD, recurrence or death was documented, up to 3 years
Population: Patients who have CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 32 | 28
months | 4.0 [1.9 to 5.7] | 3.7 [3.6 to 7.2]
Statistical Analysis 1: Comparison: Lurbinectedin vs Control (PLD or Topotecan); Duration of response between treatments; Test type: Superiority; p = 0.2631, Log Rank; Hazard Ratio (HR) = 1.406, 95% CI 2-sided [0.769 to 2.569]

7. Secondary Outcome: Duration of Response by Investigator's Assessment
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Patients who have CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 35 | 37
months | 4.3 [3.6 to 5.8] | 3.7 [3.2 to 5.6]
Statistical Analysis 1: Comparison: Lurbinectedin vs Control (PLD or Topotecan); Test type: Superiority — Duration of response between treatments; p = 0.8276, Log Rank; Hazard Ratio (HR) = 1.056, 95% CI 2-sided [0.64 to 1.743]

8. Secondary Outcome: Best Response According to Tumor Marker Evaluation (CA-125)
Description: Best response according to tumor marker evaluation (CA-125): defined as the best response obtained according to GCIG criteria. Tumor marker assessments were performed at baseline and every eight weeks from randomization until evidence of PD. Progression based on serum CA-125 levels was defined on the basis of a progressive serial elevation of serum CA-125 according to:
  A. Patients with elevated CA-125 pretreatment and normalization of CA-125 must show evidence of CA-125 greater than, or equal to, 2 times the upper limit of the reference range on 2 occasions at least 1 week apart or B. Patients with elevated CA-125 before treatment, which never normalizes, must show evidence of CA-125 greater than, or equal to, 2 times the nadir value on 2 occasions at least 1 week apart or C. Patients with CA-125 in the reference range before treatment must show evidence of CA-125 greater than, or equal to, 2 times the upper limit of the reference range on 2 occasions at least 1 week apart.
Time Frame: At baseline and every eight weeks from randomization until evidence of PD, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
Number analyzed (Participants) | 173 | 165
Participants
  Complete response | 13 | 3
  Partial response | 33 | 29
  Stable disease | 95 | 94
  Progressive disease | 17 | 16
  Unknown | 15 | 23
Statistical Analysis 1: Comparison: Lurbinectedin; ORR (%) by CA-125; Test type: Superiority; ORR (%) = 26.6, 95% CI 2-sided [20.2 to 33.8] — Percent of Participants
Statistical Analysis 2: Comparison: Control (PLD or Topotecan); ORR (%) by CA-125; Test type: Superiority; ORR (%) = 19.4, 95% CI 2-sided [13.7 to 26.3] — Percent of Participants
Statistical Analysis 3: Comparison: Lurbinectedin vs Control (PLD or Topotecan); ORR (%) by CA-125 between treatments; Test type: Superiority; p = 0.1231, Fisher Exact

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, approximately 3 years
Description: A total of 432 of 442 patients randomized in this study were treated (n=219 in the Lurbinectedin arm; n=213 in the Control arm [PLD or topotecan]) and therefore were evaluable for safety. Ten patients were not treated after randomization: two in the Lurbinectedin arm and eight in the Control arm (PLD or topotecan).
Arm/Group | Lurbinectedin | Control (PLD or Topotecan)
All-Cause Mortality (participants affected / at risk) | 170/219 | 171/213
Serious Adverse Events (participants affected / at risk) | 92/219 | 85/213
Other Adverse Events (participants affected / at risk) | 212/219 | 211/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurbinectedin (N=219) | Control (PLD or Topotecan) (N=213)
Embolism (Vascular disorders) | 2 (2) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 4 (5)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2)
Mucosal inflammation (General disorders) | 0 (0) | 3 (4)
Pain (General disorders) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorespiratory arrest (Cardiac disorders) | 3 (3) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (14) | 12 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (14) | 12 (13)
Leucopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 11 (14) | 13 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 11 (20)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 6 (6)
Ascites (Gastrointestinal disorders) | 4 (6) | 7 (11)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 24 (32) | 21 (28)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (5)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (10) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperclycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurbinectedin (N=219) | Control (PLD or Topotecan) (N=213)
Hypertension (Vascular disorders) | 12 (22) | 4 (9)
Weight decreased (Investigations) | 10 (14) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 26 (33)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (37) | 23 (34)
Anaemia (Blood and lymphatic system disorders) | 57 (155) | 77 (201)
Leucopenia (Blood and lymphatic system disorders) | 23 (39) | 21 (38)
Neutropenia (Blood and lymphatic system disorders) | 73 (167) | 89 (211)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (46) | 39 (77)
Headache (Nervous system disorders) | 26 (36) | 9 (10)
Neuropathy peripheral (Nervous system disorders) | 19 (32) | 15 (20)
Fatigue (General disorders) | 133 (328) | 113 (206)
Mucosal inflammation (General disorders) | 22 (26) | 68 (145)
Oedema (General disorders) | 25 (32) | 13 (15)
Pyrexia (General disorders) | 25 (29) | 33 (40)
Sleep disorder (Psychiatric disorders) | 22 (23) | 10 (10)
Abdominal distension (Gastrointestinal disorders) | 12 (16) | 10 (12)
Abdominal pain (Gastrointestinal disorders) | 74 (145) | 52 (73)
Ascites (Gastrointestinal disorders) | 14 (15) | 21 (43)
Constipation (Gastrointestinal disorders) | 72 (118) | 61 (84)
Diarrhoea (Gastrointestinal disorders) | 45 (71) | 35 (58)
Nausea (Gastrointestinal disorders) | 156 (390) | 92 (169)
Dyspepsia (Gastrointestinal disorders) | 14 (16) | 15 (16)
Vomiting (Gastrointestinal disorders) | 87 (196) | 58 (88)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 30 (33)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 51 (98)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 14 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (20) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (17) | 19 (22)
Decreased appetite (Metabolism and nutrition disorders) | 51 (81) | 47 (69)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (26) | 15 (28)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 20 (21)
Urinary tract infection (Infections and infestations) | 21 (25) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT02421588/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02421588/SAP_001.pdf